CLINICAL TRIAL: NCT00004255
Title: A Multi-Center, Open Label, Randomized, Active Controlled Phase II/III Clinical Trial to Evaluate the Safety and Efficacy of Processed Unrelated Bone Marrow in Patients With Acute or Chronic Leukemia
Brief Title: Treatment of Bone Marrow to Prevent Graft-Versus-Host Disease in Patients With Acute or Chronic Leukemia Undergoing Bone Marrow Transplantation
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Chimeric Therapies (Industry)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Masking: None | Purpose: Treatment
Other Study IDs: CHIMERIC-HM01; CDR0000067502 (Registry Identifier: PDQ (Physician Data Query)); WSU-10-02-99-M01-FB
Record Dates: First submitted 2000-01-28; First posted 2003-05-09 (Estimated); Last update posted 2013-07-10 (Estimated); Status verified 2002-02

CONDITIONS: Graft Versus Host Disease; Leukemia; Myelodysplastic Syndromes
Keywords: recurrent childhood acute lymphoblastic leukemia; recurrent childhood acute myeloid leukemia; recurrent adult acute myeloid leukemia; recurrent adult acute lymphoblastic leukemia; chronic phase chronic myelogenous leukemia; accelerated phase chronic myelogenous leukemia; adult acute myeloid leukemia in remission; adult acute lymphoblastic leukemia in remission; childhood acute myeloid leukemia in remission; childhood acute lymphoblastic leukemia in remission; refractory anemia with excess blasts; refractory anemia with excess blasts in transformation; secondary acute myeloid leukemia; de novo myelodysplastic syndromes; previously treated myelodysplastic syndromes; secondary myelodysplastic syndromes; graft versus host disease; childhood myelodysplastic syndromes
MeSH Terms: conditions — Graft vs Host Disease; Leukemia; Myelodysplastic Syndromes; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Acute; Leukemia, Myeloid, Chronic-Phase; Leukemia, Myeloid, Accelerated Phase; Anemia, Refractory, with Excess of Blasts | interventions — Antilymphocyte Serum; Filgrastim; Cyclophosphamide; fludarabine phosphate; Methylprednisolone; Tacrolimus; Radiotherapy

INTERVENTIONS:
Biological: anti-thymocyte globulin
Biological: filgrastim
Drug: cyclophosphamide
Drug: fludarabine phosphate
Drug: methylprednisolone
Drug: tacrolimus
Procedure: allogeneic bone marrow transplantation
Procedure: in vitro-treated bone marrow transplantation
Radiation: radiation therapy

SUMMARY:
RATIONALE: Bone marrow that has been treated to remove certain white blood cells may reduce the chance of developing graft-versus-host disease following bone marrow transplantation.

PURPOSE: Randomized phase II/III trial to compare the effectiveness of treated bone marrow with that of untreated bone marrow in preventing graft-versus-host disease in patients with acute or chronic leukemia who are undergoing bone marrow transplantation.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the efficacy of processed (cell depleted) vs unprocessed (conventional) unrelated bone marrow transplantation in reducing grade III/IV acute graft vs host disease (GVHD) in patients with acute or chronic leukemia or myelodysplastic syndromes.
* Compare the safety of these regimens in these patients.
* Compare the disease-free survival rate at 100 days and at 6 months in patients treated with these regimens.
* Compare the time to engraftment and percent engraftment in patients treated with these regimens.
* Compare the reduction rate of grade II or greater acute and chronic GVHD in patients treated with these regimens.

OUTLINE: This is a randomized, open-label, multicenter study. Patients are stratified according to degree of HLA matching and disease (chronic vs acute). Acute myelogenous leukemia patients are further stratified according to prior myelodysplastic syndromes (yes vs no). Patients are randomized to one of two bone marrow transplantation arms.

All patients receive a conditioning regimen comprising fludarabine IV on day -6, cyclophosphamide IV on days -5 and -4, anti-thymocyte globulin IV on days -4 and -2, and total body irradiation on days -3 to 0. Patients also receive methylprednisolone IV every 12 hours for 4 doses on days -2 to 0. Tacrolimus IV is administered continuously on day -1 and continues either orally or IV for 6 months. Bone marrow is infused on day 0. Filgrastim (G-CSF) is administered subcutaneously from day 0 until blood counts recover.

* Arm I: Patients receive allogeneic bone marrow that has been processed to produce a mononuclear cell preparation.
* Arm II: Patients receive unprocessed allogeneic bone marrow. Patients are followed weekly for 100 days and then at 6 months.

PROJECTED ACCRUAL: A total of 260 patients will be accrued for this study within 17 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of one of the following:

  * Acute myelogenous leukemia (AML) or acute lymphocytic leukemia (ALL) in first early relapse, second remission, or subsequent remission
  * AML in first complete remission with one of the following adverse features:

    * Antecedent hematologic disorder such as myelodysplasia
    * AML resulting from prior chemotherapy or radiotherapy
    * More than 1 course of induction chemotherapy to achieve remission or adverse cytogenetics such as Philadelphia chromosome 9:22, +8, +11; abnormal 12p; or deletions of chromosomes 5, 7, or 20 (3:3)
  * ALL in first complete remission with poor risk cytogenetics such as

    * Philadelphia chromosome 9:22, 8:14, or 4:11 OR
    * WBC greater than 100,000/mm3 OR
    * Time to achieve complete remission more than 4 weeks
  * Chronic myelogenous leukemia in chronic or accelerated phase
  * Myelodysplastic syndromes

    * Refractory anemia with excess blasts (RAEB) OR
    * RAEB in transformation
* Unrelated bone marrow donor available

  * If matched at 6 of 6 HLA-A, -B, and -DR loci, patient must be 12 to 50 years
  * If matched at 5 of 6 loci, patient must be 12 to 35 years
* No matched sibling donor available
* No uncontrolled CNS leukemia

PATIENT CHARACTERISTICS:

Age:

* See Disease Characteristics
* 12 to 50

Performance status:

* Karnofsky 70-100%

Life expectancy:

* At least 12 weeks

Hematopoietic:

* See Disease Characteristics

Hepatic:

* Bilirubin less than 2.5 times upper limit of normal (ULN)
* SGOT or SGPT less than 2.5 times ULN

Renal:

* Creatinine no greater than 1.5 mg/dL

Cardiovascular:

* LVEF greater than 50% without medication

Pulmonary:

* DLCO and FVC at least 50% predicted

Other:

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No other serious medical illness
* No uncontrolled diabetes mellitus
* No uncontrolled and/or active infection
* HIV negative

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* At least 3 weeks since prior immunotherapy and recovered
* At least 1 year since prior autologous transplantation
* No prior allogeneic transplantation

Chemotherapy:

* See Disease Characteristics
* At least 3 weeks since prior chemotherapy (except hydroxyurea) and recovered

Endocrine therapy:

* At least 3 weeks since prior hormonal therapy and recovered

Radiotherapy:

* See Disease Characteristics
* At least 3 weeks since prior radiotherapy and recovered
* No prior radiotherapy at doses that would preclude study

Surgery:

* Not specified

Ages: 12 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Dates: Start 2000-03; Study Completion 2003-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James N. Lowder, MD, Study Chair — Chimeric Therapies
Locations (15):
- United States (15):
  - University of California San Diego Cancer Center, La Jolla, California
  - Presbyterian-St Luke's Medical Center, Denver, Colorado
  - Lombardi Cancer Center, Washington D.C., District of Columbia
  - Shands Hospital and Clinics, University of Florida, Gainesville, Florida
  - Indiana Blood and Marrow Transplantation, Indianapolis, Indiana
  - James Graham Brown Cancer Center, Louisville, Kentucky
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - University of Rochester Cancer Center, Rochester, New York
  - New York Medical College, Valhalla, New York
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Oregon Cancer Center, Portland, Oregon
  - Hahnemann University Hospital, Philadelphia, Pennsylvania
  - University of Texas - MD Anderson Cancer Center, Houston, Texas
  - South Texas Cancer Institute, San Antonio, Texas
  - Massey Cancer Center, Richmond, Virginia